CLINICAL TRIAL: NCT01082198
Title: Adjuvant Vaccination With Melanoma Antigen Pulsed Dendritic Cells (DCs) in Stage III Melanoma Patients
Brief Title: Melanoma Vaccine in Treating Patients With Stage III Melanoma After Surgery to Remove Lymph Nodes
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000666511; MSCMI-21/01/02; EU-21006
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2010-03

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma
MeSH Terms: conditions — Melanoma | interventions — Flow Cytometry; Chemotherapy, Adjuvant

INTERVENTIONS:
Biological: HLA-A1-binding MAGE-1/MAGE-3 multipeptide-pulsed autologous dendritic cell vaccine
Biological: HLA-A2-binding TYR/MART-1/gp100 multipeptide-pulsed autologous dendritic cell vaccine
Biological: autologous melanoma lysate-pulsed autologous dendritic cell vaccine
Biological: autologous melanoma lysate/KLH-pulsed autologous dendritic cell vaccine
Biological: dendritic cell-idiotype-keyhole limpet hemocyanin vaccine
Other: flow cytometry
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Vaccines made from dendritic cells and tumor antigen peptides or a person's tumor cells may help the body build an effective immune response to kill tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best way to give melanoma vaccine in treating patients with stage III melanoma after surgery to remove the lymph nodes.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of adjuvant melanoma vaccine comprising autologous dendritic cells pulsed with tumor antigen peptides in patients with stage III melanoma following lymphadenectomy.
* Determine the immune response (skin test of delayed-type hypersensitivity and flow cytometric enumeration of peripheral blood CD8+ lymphocytes producing IFN-γ) to this regimen in these patients.
* Determine clinical outcome (disease-free survival, overall survival, and adverse events) in patients treated with this regimen.

OUTLINE: Patients undergo leukapheresis for collection of peripheral blood mononuclear cells (PBMCs) and bone marrow mononuclear cells. Autologous dendritic cells (DCs) prepared from PBMCs and bone marrow mononuclear cells are exposed to various antigens and peptides, and autologous tumor cell lysate, if available. Patients receive autologous DCs pulsed with melanoma-associated antigen peptides, and autologous DCs pulsed with tumor lysates (if available), subcutaneously in weeks 0, 2, 5, 8, 12, 16, 20, 26, 31, 50, and 102. Patients with no evidence of disease may receive another booster injection 5 years after the start of vaccination.

Blood samples are examined via flow cytometry and skin testing is performed to evaluate immune response.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage III melanoma

  * Has undergone therapeutic lymphadenectomy
  * More than 1 lymph node involvement or extracapsular extension of metastatic melanoma cells (stage N1b-N3 disease according to AJCC 2002)
* HLA type A1 and/or A2 or A3 (if autologous tumor lysate is available)
* No presence of distant metastases

PATIENT CHARACTERISTICS:

* No other malignancy
* No evidence of lung, heart, liver, or renal failure or severe neurologic disorder
* No autoimmune disease or atopic allergy
* No HIV infection or presence of anti-HIV antibodies
* No presence of hepatitis B surface antigen or antibodies against hepatitis C virus

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2002-10; Primary Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Immune response
Disease-free survival
Overall survival
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Sergiusz Markowicz, MD, Principal Investigator — Maria Sklodowska-Curie National Research Institute of Oncology
Locations (1):
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology - Warsaw, Warsaw, Poland